# Plication of Fascia Transversalis and Its Role in Reduction of Seroma Formation Post Laparoscopic Transabdominal Preperitoneal Repair of Direct Inguinal Hernia

Patient Information and Consent Form

Ву

Dr. Mohammed Elshwadfy Nageeb Abdelaziz

Ethical Approval Number: MS 204-2024

Faculty of Medicine Cairo University 2025

#### Patient Information and Consent Form

## Study Title:

Plication of Fascia Transversalis and Its Role in Reduction of Seroma Formation Post Laparoscopic Transabdominal Preperitoneal Repair of Direct Inguinal Hernia

# Purpose of the Study:

You are invited to take part in this study, which aims to see if tightening a thin layer of tissue (fascia transversalis) during hernia surgery helps reduce fluid collection (seroma) after the operation.

# What Will Happen to You:

- You will undergo standard laparoscopic hernia repair (TAPP).
- In some patients, an extra step of tightening the fascia will be added.
- You will be followed up after surgery with routine visits and ultrasound.

## Possible Benefits:

- Better healing after surgery.
- Less chance of fluid collection.

#### Possible Risks:

- Temporary pain or discomfort at the surgery site.
- Rare risks such as bleeding, infection, or recurrence of hernia.
- Risks will not be more than standard hernia surgery.

## Confidentiality:

Your information will be kept private. Your name will not appear in any report or publication.

# Voluntary Participation:

Joining the study is your choice. You can refuse or stop at any time without affecting your treatment.

# Contact:

If you have any questions, please contact your doctor or the research team.

## Consent Statement:

I have read and understood this information. I agree to participate in this study.

| Patient ' | s Name: |
|-----------|---------|
| Signatur | e: |
| Date: | |